CLINICAL TRIAL: NCT02452216
Title: MR Imaging of Inflammatory Responses in the Central Nervous System With Ferumoxytol-Enhanced MRI
Brief Title: Using Ferumoxytol-Enhanced MRI to Measure Inflammation in Patients With Brain Tumors or Other Conditions of the CNS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Michael Iv (Other)
Responsible Party: Sponsor-Investigator, Michael Iv, Clinical Assistant Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BRNCNS0007; NCI-2015-00435 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 26570 (Other: Stanford IRB)
Record Dates: First submitted 2015-05-20; First posted 2015-05-22 (Estimated); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Brain Injury; Central Nervous System Degenerative Disorder; Central Nervous System Infectious Disorder; Central Nervous System Vascular Malformation; Hemorrhagic Cerebrovascular Accident; Ischemic Cerebrovascular Accident; Primary Brain Neoplasm; Brain Cancer; Brain Tumors
MeSH Terms: conditions — Brain Injuries; Neurodegenerative Diseases; Central Nervous System Infections; Central Nervous System Vascular Malformations; Hemorrhagic Stroke; Ischemic Stroke; Brain Neoplasms | interventions — Ferrosoferric Oxide; Tissue Array Analysis; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ferumoxytol group (Experimental): All subjects in the experimental arm will have a single intravenous dose of ferumoxytol (5 mg Fe/kg), to be administered 24 hours before the subject undergoes ferumoxytol-enhanced magnetic resonance imaging (MRI). These subjects will subsequently undergo surgery, and tissue analysis of surgically resected samples (specifically the number of iron-containing and non-iron-containing macrophages) will be correlated with imaging features on ferumoxytol-enhanced MRI.
  Interventions: Drug: Ferumoxytol; Other: Tissue Analysis; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Drug: Ferumoxytol — Undergo ferumoxytol-enhanced MRI
  Other Names: Feraheme; FERUMOXYTOL NON-STOICHIOMETRIC MAGNETITE
Other: Tissue Analysis — Correlative analysis for macrophage detection and quantification. This applies for all patients in the experimental arm who undergo ferumoxytol infusion.
Procedure: Magnetic Resonance Imaging — All subjects in the experimental arm who undergo ferumoxytol infusion will subsequently have MRI.
  Other Names: Magnetic Resonance Imaging Scan; MRI

SUMMARY:
This pilot clinical trial study will assess the inflammatory response of brain tumors or other central nervous system conditions in pediatric and adult patients using ferumoxytol-enhanced MRI. Imaging features will be correlated with the number of inflammatory cells (macrophages) at histopathology. Determining the extent of inflammation associated with pathologies in the central nervous system may be helpful for diagnostic and prognostic purposes as well as monitoring treatment response of current and future immunotherapies.

DETAILED DESCRIPTION:
In this study, we will establish the MR imaging characteristics of macrophages in malignant brain tumors and other CNS conditions in the pediatric and adult populations using ferumoxytol, an ultrasmall superparamagnetic iron oxide (USPIO) particle that is approved for the treatment of iron deficiency anemia in patients with chronic kidney disease. The investigators will correlate the MR signal of ferumoxytol uptake with the number of macrophages in surgical specimen at histopathology. This information may potentially offer clinicians a new means for risk stratification and monitoring treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with suspected brain tumor diagnosed by MRI
* Patients undergoing neuro-imaging evaluation by the neurosurgical service for other indications (e.g. vascular malformations, traumatic brain injury, ischemic and hemorrhagic stroke, CNS infections, and neuro-degenerative diseases)

Exclusion Criteria:

* Informed consent cannot be obtained either from the patient or legal representative
* Severe coexisting or terminal systemic disease that limits life expectancy or that may interfere with the conduct of the study
* Contraindication to MRI (metal implants)
* Hemosiderosis/hemochromatosis
* Need for sedation or anesthesia (claustrophobia) that will not otherwise be undertaken as part of routine clinical care (e.g. routine MRI under sedation already planned)
* Known hypersensitivity to Feraheme (ferumoxytol) or any of its components
* Iron overload from any cause (not just hemosiderosis or hemochromatosis), even if secondary to frequent blood transfusions, severe chronic hemolysis, excess dietary or parenteral iron, or any other etiology

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-06-10 (Actual); Primary Completion 2017-01-12 (Actual); Study Completion 2017-01-12 (Actual)

PRIMARY OUTCOMES:
Obtain measurements of iron concentration (indicative of ferumoxytol uptake) on T2*-weighted MR images. | Day 1

SECONDARY OUTCOMES:
Determine the number of macrophages in resected/biopsied samples at histopathology. | Days 2-4

CONTACTS AND LOCATIONS:
Overall Officials: Michael Iv, MD, Principal Investigator — Stanford University Hospitals and Clinics
Locations (1):
- Stanford University Hospitals and Clinics, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No